CLINICAL TRIAL: NCT01462994
Title: Prospective, Explorative Trial for the Detection of Circulating Cell-free Tumor DNA in the Plasma of Patients With Gastrointestinal Stromal Tumors (GIST)Harboring Activating Mutations of CKIT or PDGFRA Pre/Post Surgery or Pre/Under Treatment With a Tyrosine Kinase Inhibitor or Progressive Disease Irrespective of Current or Planned Treatment. An Open-label, Non-randomized, Multicenter Phase IIIb Clinical Trial
Brief Title: Detection of CF-DNA in Patients With Gastrointestinal Stromal Tumors (GIST)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CSTI571BDE78T
Record Dates: First submitted 2011-10-25; First posted 2011-11-01 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Patients with GIST treated with standard therapy harboring activating mutations of CKIT and PDGFRA
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (No Intervention)
  Interventions: Other: Blood will be withdrawn at baseline and in intervals of 3 months for a total period of 2 years

INTERVENTIONS:
Other: Blood will be withdrawn at baseline and in intervals of 3 months for a total period of 2 years

SUMMARY:
Activating mutations of the kinases CKIT or PDGFRA can be detected in 90% of cases by DNA sequence analysis of a pathological specimen. These mutated genomic DNA fragments are highly specific for the tumor and are released by the tumor into the circulation. Allele-specific PCR can be used to specifically amplify and quantify mutated CKIT and PDGFR DNA fragments.

The current trial aims to evaluate whether tumor DNA carrying mutations for CKIT and PDGFRA can be detected and quantified in the plasma of patients with active GIST, and whether detection can be correlated with the clinical course of disease either under therapy or in progressive disease irrespective of current therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male or female patients aged >= 18 years
* Histologically confirmed GIST
* Known activating mutation of CKIT or PDGFRA and tissue sample can be provided for central mutation analysis or mutation status unknown and tissue sample can be provided for central mutation analysis at baseline
* Routinely planned follow-up visits in no longer than three months intervals (+ 14 days) including local standard of care diagnostic imaging (CT, PET- CT, or MRI)
* At least one GIST lesion that can be measured by CT, PET-CT, or MRI
* Planned surgery of one or more disease manifestations or planned TKI treatment (such as imatinib or sunitinib) in neoadjuvant or palliative intention or disease progression irrespective of current/planned treatment
* Life expectancy of at least three months

Exclusion Criteria:

* Wild type sequence for CKIT exon 9, 11, 13, 14, 17, 18 and PDGFRA exon 18
* Tissue sample can not be provided for central mutation analysis
* Surgery of primary or progressive lesions already completed and currently no evidence of progressive lesions
* Patients currently receiving adjuvant TKI treatment after surgery and no evidence of progressive lesions
* Patients currently receiving palliative TKI treatment and no evidence of progressive lesions
* Planned follow-up intervals including CT, PET-CT or MRI at more than three months intervals (+ 14 days)
* Coexisting medical condition or treatment that could interfere with the ability of the patient to comply with planned treatment interventions (surgery or TKI treatment) or regular follow-up visits
* Patients unwilling to or unable to comply with the planned therapeutic intervention (surgery or TKI treatment) or to comply with the regular follow-up visits including blood sample collection
* Pregnancy and lactation
* Presence of chronic inflammatory diseases, autoimmune diseases, or liver cirrhosis
* Known HIV and/or hepatitis B or C infection
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix and basal or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-11; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with histologically proven GIST, measurable lesion in imaging and activating CKIT and PDGFRA mutation, where detection of tumor specific DNA encoding for mutated CKIT or PDGFA is possible in the plasma at least at one timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Nikolas von Bubnoff, PD Dr., Study Chair — Klinikum rechts der Isar
Locations (1):
- Klinikum rechts der Isar - III. Medizinische Klinik und Poliklinik, Munich, Bavaria, Germany